CLINICAL TRIAL: NCT03172936
Title: A Phase Ib, Open Label, Multicenter Study of the Safety and Efficacy of MIW815 (ADU-S100) Administered by Intratumoral Injection With PDR001 to Patients With Advanced/Metastatic Solid Tumors or Lymphomas
Brief Title: Study of the Safety and Efficacy of MIW815 With PDR001 in Patients With Advanced/Metastatic Solid Tumors or Lymphomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMIW815X2102J; 2017-000707-25 (EudraCT Number)
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Solid Tumors and Lymphomas
Keywords: injected lesion; distal lesion; abscopal activity; intratumoral; checkpoint inhibitor; cyclic dinucleotide; programmed cell death
MeSH Terms: conditions — Lymphoma | interventions — spartalizumab

STUDY DESIGN:
Intervention Model Description: The study was comprised of two treatment arms.
  Group A included patients with accessible solid tumors and lymphomas. This group received a fixed dose of PDR001 intravenous on day 1 of every 28 day cycle and intratumoral injections of MIW815 (ADU-S100) on days 1, 8 and 15 of every 28 day cycle.
  Group B included patients with accessible solid tumors and lymphomas. This group received a fixed dose of PDR001 intravenous on day 1 of every 28 day cycle and an intratumoral injection of MIW815 (ADU-S100) on day 1 of every 28 day cycle.
  Once the maximum tolerated dose and/or recommended dose for expansion had been determined, the plan was to open the expansion part of the study. However, the dose expansion phase of the study was not opened to enrollment due to the program's early termination.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dosing Schedule A (Experimental): Patients were treated with MIW815 (ADU-S100) via intratumoral injection for 3 weeks followed by one week off in combination with a fixed intravenous dose of PDR001 given once per month
  Interventions: Drug: MIW815; Biological: PDR001
- Dosing Schedule B (Experimental): Patients were treated with MIW815 (ADU-S100) via intratumoral injection given once a month in combination with a fixed intravenous dose of PDR001 given once per month
  Interventions: Drug: MIW815; Biological: PDR001

INTERVENTIONS:
Drug: MIW815 — MIW 815 (ADU-S100) is a STING agonist
Biological: PDR001 — PDR001 is an anti-PD-1 antibody

SUMMARY:
The purpose of this study was to characterize the safety, tolerability, pharmacokinetics, pharmacodynamics and antitumor activity of MIW815 (ADU-S100) in combination with PDR001.

DETAILED DESCRIPTION:
This was a Phase Ib, multi-center, open-label study to characterize the safety, tolerability, pharmacokinetics, pharmacodynamics and preliminary antitumor activity of MIW815(ADU-S100) in combination with the PD-1 checkpoint inhibitor PDR001. Two different schedules were explored in two dose escalation groups in accessible cutaneous or subcutaneous lesions. The optional dose confirmation group exploring intratumoral injection of viscerally located lesions was not opened due to the program's early termination.

Group A included patients with accessible solid tumors and lymphomas. This group received a fixed dose of PDR001 i.v. on day 1 of every 28 day cycle and intratumoral injections of MIW815 (ADU-S100) on days 1, 8 and 15 of every 28 day cycle. Group B included patients with accessible solid tumors and lymphomas. This group received a fixed dose of PDR001 i.v. on day 1 of every 28 day cycle and an intratumoral injection of MIW815 (ADU-S100) on day 1 of every 28 day cycle.

Once the dose and dose schedule had been confirmed, the plan was to open the dose expansion part of the study. However, the expansion phase of the study was not opened to enrollment due to the program's early termination.

ELIGIBILITY:
Inclusion Criteria:

ECOG ≤ 1 Willing to undergo tumor biopsies from injected and distal lesions

Must have two biopsy accessible lesions:

Exclusion Criteria:

Symptomatic or untreated leptomeningeal disease. Presence of symptomatic central nervous system metastases Impaired cardiac function or clinically significant cardiac disease Active autoimmune disease or a documented history of autoimmune disease, except vitiligo or resolved childhood asthma/atopy.

Active infection requiring systemic antibiotic therapy. Known history of human immunodeficiency virus infection. Active Epstein-Barr virus, hepatitis B virus or hepatitis C virus Malignant disease, other than that being treated in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | 24 months
  A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first cycle of treatment with the combination of MIW815 (ADU-S100) and PDR001

SECONDARY OUTCOMES:
AUC inf | 36 months
  The area under the concentration-time curve extrapolated to infinity (mass*time/volume)
AUC last | 36 months
  The area under the concentration (AUC) -time curve calculated to the last quantifiable concentration point (mass* time/volume)
AUC tau | 36 months
  Area under the concentration-time curve calculated to the end of the dosing interval (tau) (mass* time/volume)
Tmax | 36 months
  The time to reach the maximum observed concentration (time)
Cmax | 36 months
  The maximum observed concentration (Cmax) following dose administration (mass/volume)
Lambda_z | 36 months
  Terminal elimination rate constant (1/time)
CL/F | 36 months
  Apparent systemic clearance of drug from the plasma (volume x time -1)
T1/2 | 36 months
  Elimination half-life, determined as 0.693/Lambda_z (time)
Vz/F | 36 months
  Apparent volume of distribution during the terminal elimination phase (volume)
Best overall response (BOR) | 36 months
  Best overall response will be summarized
Overall response rate (ORR) | 36 months
  Overall response rate will be summarized with accompanying 90% exact binomial confidence interval (CI).
Progression free survival (PFS) | 36 months
  The survival function will be estimated using the Kaplan-Meier product limit method. Median duration, with a two-sided Brookmeyer-Crowley 90% confidence interval and Kaplan-Meier estimates of survival proportions will be provided at specified time points.
Disease control rate (DCR) | 36 months
  The disease control rate is calculated as the percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease
Time to response (TTR) | 36 months
  Time To Response is the time from first dose to first documented response (CR or PR). TTR will be summarized
Duration of Response (DOR) | 36 months
  Duration of response is defined as the time from the date of the first documented response (CR or PR), to the date of first documented progression, or death due to study indication. Estimates will use Kaplan-Meier method
Tumor infiltrating lymphocytes (TIL) | 36 months
  Induction of TILs in the injected lesion (local PD effect) and in a non-injected lesion (distal PD effect) will be assessed using paired tumor samples at screening and on-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lewis, MD, Study Director — Novartis
Locations (12):
- United States (4):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Novartis Investigative Site, Chicago, Illinois
  - MD Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (2):
  - Novartis Investigative Site, North Sydney, New South Wales
  - Novartis Investigative Site, Melbourne, Victoria
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Essen, Germany
- Novartis Investigative Site, Chuo Ku, Tokyo, Japan
- Novartis Investigative Site, Amsterdam, Netherlands
- Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia, Spain
- Novartis Investigative Site, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gogoi H, Mansouri S, Jin L. The Age of Cyclic Dinucleotide Vaccine Adjuvants. Vaccines (Basel). 2020 Aug 13;8(3):453. doi: 10.3390/vaccines8030453. PMID 32823563
- See also: Study Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17869
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=987